CLINICAL TRIAL: NCT02695901
Title: Anti-plaque Effect of 0.12% Chlorhexidine Gluconate Rinsing and Nanoparticle Solution of 0.3% Melaleuca Alternifolia: A Randomized Crossover Clinical Trial
Brief Title: Effect of Different Mouthrinses in Plaque Formation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Collaborators: Centro Universitário Franciscano (Unknown)
Responsible Party: Principal Investigator, Maísa Casarin, MsC, Federal University of Santa Maria, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 52275816.0.0000.5346; 1.399.643 (Other: Ethics Committee in Research)
Record Dates: First submitted 2016-02-21; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Dental Plaque
Keywords: Plaque index; Melaleuca alternifolia oil.; Nanoparticles
MeSH Terms: conditions — Dental Plaque | interventions — chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Chlorhexidine gluconate (0,12%) (Experimental): Subjects will rinse twice daily with 15 ml mouthrinse containing Chlorhexidine gluconate (0.12%).
  Interventions: Drug: Chlorhexidine gluconate 0.12% (PerioGard®)
- M. alternifolia oil (Nanoparticle solution) (Experimental): Subjects will rinse twice daily with 15 ml mouthrinse containing nanoparticles of M. alternifolia oil (0.3%).
  Interventions: Drug: Nanoparticle solution of M. alternifolia oil (0.3%).

INTERVENTIONS:
Drug: Chlorhexidine gluconate 0.12% (PerioGard®) — At baseline, subjects will receive a professional prophylaxis and will be instructed to withdrawal oral hygiene methods for 3 days. At day 4, 2 contra-lateral quadrants will be randomly chosen to receive a professional prophylaxis, being controls for plaque-covered surfaces. Subjects will then start to rinse twice daily with 15 ml mouthrinse containing Chlorhexidine gluconate (0.12%). Plaque indices will be recorded at baseline, day 4, and day 7.
  Arms: Chlorhexidine gluconate (0,12%)
Drug: Nanoparticle solution of M. alternifolia oil (0.3%). — At baseline, subjects will receive a professional prophylaxis and will be instructed to withdrawal oral hygiene methods for 3 days. At day 4, 2 contra-lateral quadrants will be randomly chosen to receive a professional prophylaxis, being controls for plaque-covered surfaces. Subjects will then start to rinse twice daily with 15 ml mouthrinse containing a nanoparticle solution of M. alternifolia oil (0.3%). Plaque indices will be recorded at baseline, day 4, and day 7.
  Arms: M. alternifolia oil (Nanoparticle solution)

SUMMARY:
Although several studies have assessed the efficacy of chlorhexidine in treating gingivitis and reducing biofilm formation, the side effects of a long-term use are unpleasant for patients. Melaleuca alternifolia oil has been considered as an alternative because of its anti-inflammatory properties. However, little is know about the efficacy of its nanoparticles. The purpose of this study is to compare the effect of 0.12% chlorhexidine (Periogard ®) and a nanoparticle solution of 0.3% M. alternifolia oil in reducing biofilm formation in plaque-free and plaque-covered teeth surfaces.

DETAILED DESCRIPTION:
This will be a randomized crossover clinical trial, double blind, in which individuals will be randomly assigned into two different treatments: daily mouthrinse of chlorhexidine gluconate (0.12%) or daily mouthrinse of a nanoparticle solution of M. alternifolia (0.3%) during a period of oral hygiene withdrawal.

The test panel will consist of 59 students from the Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil. All subjects will receive written and oral explanations regarding the purpose and design of this study. Those who met the inclusion criteria will be selected for a dental screening appointment, being removed in the presence of any exclusion criteria. All volunteers will be asked to sign an informed consent before the experimental period.

The following clinical parameters will be assessed:

* Plaque index (PI) Quigley and Hein modified by Turesky.
* Gingival crevicular fluid (GCF) will be measured with an electronic gingival fluid measuring device (Periotron®).
* Gingival abrasion (GA) using 2-Tone disclosing solution.
* Perception of appreciation (Questionnaire-VAS scale). Descriptive analysis of PI data will be performed using averages, standard deviations and average percentage of sites with different PI scores. The normal distribution of the data will be evaluated by the Kolmogorov-Smirnov test. Analysis of variance (ANOVA) with repeated measures will be used to test for differences between groups. Paired student's t-test will be conducted to test whether there were significant differences between the baseline measurements of PI, GA, GCF and perception of appreciation after the use of mouthwash. The statistical tests will be performed using the program SPSS 20.0 (Statistical Package for the Social Sciences, Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be systemically healthy;
* Must have at least six teeth per quadrant;
* Must not be undergoing medical treatment;

Exclusion Criteria:

* Allergies or hypersensitivity to the components (Chlorhexidine Gluconate or M. alternifolia oil nanoparticles);
* Antibiotic therapy within 3 months prior to baseline examination;
* History of periodontal disease;
* Marginal bleeding index higher than 15%;
* Oral mucosal lesions;
* Pregnancy or breastfeeding;
* Presence of active infectious foci (endodontic abscesses);
* Presence of plaque retentive factors (caries, aesthetic or ill-fitting restorations, orthodontic appliances, fixed or removable prosthesis);
* Smokers;
* Systemic conditions (diabetes, immunosuppression);
* Use of any mouthwash within 21 days prior to baseline examination;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Dental plaque/biofilm formation. | 7 days.

SECONDARY OUTCOMES:
Gingival abrasion. | 7 days.

OTHER OUTCOMES:
Gingival crevicular fluid- measured through an electronic gingival fluid measuring device (Periotron®) | 7 days.
  The volume of gingival fluid will be measured at two locations per quadrant.
Perception of appreciation- questionnaire | 7 days.
  Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio B. Zanatta, PhD, Study Director — Adjunct Professor

REFERENCES:
- [Background] Rahman B, Alkawas S, Al Zubaidi EA, Adel OI, Hawas N. Comparative antiplaque and antigingivitis effectiveness of tea tree oil mouthwash and a cetylpyridinium chloride mouthwash: A randomized controlled crossover study. Contemp Clin Dent. 2014 Oct;5(4):466-70. doi: 10.4103/0976-237X.142813. PMID 25395761